CLINICAL TRIAL: NCT03940170
Title: Clinical Effectiveness of Quantitative Light Fluorescence Based Device (Vistacam Proof) in Comparison With ICDAS-II and Histological Validation in Detection of Initial Pits and Fissures Caries:: Diagnostic Accuracy Study
Brief Title: Clinical Effectiveness of(VistaProof)in Comparison With ICDAS-II & Histological Validation for Detecting Occlusal Caries
Status: Completed | Type: Observational
Sponsor: Mohamed samy El-sayed (Other)
Responsible Party: Sponsor-Investigator, Mohamed samy El-sayed, assistant lecturer, Cairo University
Organization: Cairo University (Other)
Other Study IDs: 2222
Record Dates: First submitted 2019-04-25; First posted 2019-05-07 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Light Fluorescence Device

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- vistacam
  Interventions: Device: vistacam proof
- ICDAS II
  Interventions: Other: ICDASII
- Fissurotomy
  Interventions: Device: vistacam proof; Other: ICDASII; Procedure: fissurotomy

INTERVENTIONS:
Device: vistacam proof — Light fluorescence device
  Groups: Fissurotomy; vistacam
Other: ICDASII — visual examination
  Groups: Fissurotomy; ICDAS II
Procedure: fissurotomy — histological validation
  Groups: Fissurotomy

SUMMARY:
a diagnostic accuracy study control trial is to be held to evaluate the Clinical performance of quantitative light fluorescence based device (Vistacam Proof) in comparison with the visual examination and histological validation in detection of initial pits and fissures caries

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 15 to 50 years.
* Patient at least has one posterior pits and fissure occlusal caries.
* No gender restriction
* Co-operative patients who signed the informed consent.
* Good general health
* Acceptable oral health

Exclusion Criteria:

* Pregnancy.
* Disabilities.
* Systemic disease or severe medical complications.
* Allergic history concerning methacrylate.
* Rampant caries.

Ages: 15 Years to 50 Years | Sex: All
Age Groups: Child, Adult
Study Population: Egyptian population
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-08-09 (Actual)

PRIMARY OUTCOMES:
pits and fissure caries | through study completion, an average of 1 year
  occlusal pits and fissure caries in posterior teeth non-cavitated

CONTACTS AND LOCATIONS:
Locations (1):
- The British University in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided